CLINICAL TRIAL: NCT04547179
Title: Medicinal vs. Orthotic Comparison for Migraine Prevention: A Double-Blind Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Manhattan Beach Orthodontics (Other)
Responsible Party: Principal Investigator, Dr. Sunitha Bharadia, Principal Investigator, Manhattan Beach Orthodontics
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0001
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Migraine
Keywords: Migraine; Ajovy; facial exercise; fremanezumab-vfrm
MeSH Terms: conditions — Migraine Disorders | interventions — erenumab; Sodium Chloride; Salts

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- BLAfit® usage (Experimental): In this arm, subjects will used the fixed orthotic device called BLAfit® for one minute of facial exercise a day for three months.
  Interventions: Device: BLAfit®
- fremanezumab-vfrm (Experimental): Subjects in this arm will receive three Ajovy® (fremanezumab-vfrm) injections at the start of month 2. This will be conducted in a double-blind fashion, as both the clinician providing the injection, and the subject, will not know if the injection is actually Ajovy® or just saline.
  Interventions: Drug: Fremanezumab-Vfrm
- Saline injection (Placebo Comparator): This is a placebo that is used to counter Arm #2- the Ajovy® injections. Subjects in this arm will receive three saline injections at the start of month 2 that will mimic the Ajovy® injections. This will be conducted in a double-blind fashion, as both the clinician providing the injection, and the subject, will not know if the injection is actually Ajovy® or just saline.
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Fremanezumab-Vfrm — Patients will receive three injections of Ajovy® if in the corresponding arm of the study.
  Other Names: Ajovy®
  Arms: fremanezumab-vfrm
Device: BLAfit® — Usage of the BLAfit device, a fixed orthotic appliance that allows users to tone facial muscles with one minute usage per day
  Other Names: Bella Lip Appliance®; BLA®
  Arms: BLAfit® usage
Other: Saline — Patients will receive three injections of saline if in the corresponding arm of the study. This is a placebo meant to simulate the Ajovy® injection.
  Other Names: salt and water solution
  Arms: Saline injection

SUMMARY:
To understand the impacts of using a fixed orthotic facial exercise appliance (BLAfit®) for migraine reduction, as compared to medication (fremanezumab-vfrm) and control.

DETAILED DESCRIPTION:
The investigators will be studying the impacts of using an orthotic facial exercise device (BLAfit®) in the prevention of migraines for those who suffer from roughly 10-15 migraines per month. In order to test the efficacy of this device and its exercise routine, investigators will have one arm of our study receive the BLAfit® device and perform the exercises for one minute daily for three months. In Arm #2, there will be another treatment: Ajovy® (fremanezumab-vfrm) injections- which is a known and commonly practiced clinical prevention treatment for migraine patients. Patients in this arm will receive three injections of Ajovy, which is will be meant to last 3 months. In addition, investigators will have a placebo group that will receive three saline injections, which are meant to mimic the three Ajovy® injections. Arms #2 and #3 of this study will be conducted in a double-blind fashion, as both the clinician providing the injections and the patients receiving the injections will not know if the injecting substance is Ajovy or saline, so as to minimize bias. All patients in all three months will log their number and pain level of their migraines each day for three months. Upon conclusion, they will meet with our in-house neurologist (Principal Investigator & Sponsor) for a final in-person evaluation and questionnaire. Results from the three groups will then be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Those eligible to participate must be between the ages of 18 to 55 years.
* The individual must experience at least 2 migraines per week.
* They must be capable of visiting the medical facility in Manhattan Beach, California where the in-person screening and final evaluation will be conducted (following COVID-19 public health guidelines).
* They must be able to communicate with the study team via any teleconferencing service such as Zoom, Google Hangouts, or FaceTime.

Exclusion Criteria:

* Patients must not have any intracranial pathology, neurological or psychological conditions, epilepsy, cancer, any history of chemotherapy, hospitalized for depression, psychiatric conditions, seizures, or tumors.
* Patients cannot have taken Botox® for migraine treatments.
* Patients cannot have had a history of head or neck surgery.
* Patients cannot be taking: propranolol, amitriptyline, flunarizine, topiramate, combination, galcanezumab-gnlm, fremanezumab-vfrm, or erenumab-aooe.
* Patients must not be deemed a vulnerable subject (including but not limited to: children, prisoners, pregnant women, mentally disabled persons).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-04-15 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Frequency and Pain Level of Migraines Post-Treatment | 4 months after start
  The frequency and pain level of subjects' migraines will be assessed upon the conclusion of the study through surveying and comparing to previous survey data.

CONTACTS AND LOCATIONS:
Overall Officials: Sunitha Bharadia, MD, Principal Investigator — Manhattan Beach Orthodontics
Locations (1):
- Manhattan Beach Orthodontics, Manhattan Beach, California, United States

IPD SHARING:
Plan to Share IPD: No